CLINICAL TRIAL: NCT06980142
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating CM512 Injection in Subjects With Moderate-to-Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Study of CM512 in Subjects With Moderate-to-Severe Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM512-104101
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental)
  Interventions: Biological: CM512
- Dose 2 (Experimental)
  Interventions: Biological: CM512
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CM512 — Administered SC
  Arms: Dose 1; Dose 2
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
A Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase II Study to Explore the Efficacy and Safety of CM512 Injection in Adults with Moderate-to-Severe Chronic Obstructive Pulmonary Disease (COPD)

DETAILED DESCRIPTION:
This is a Phase II, multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the safety and efficacy of CM512 in adults with moderate-to-severe chronic obstructive pulmonary disease (COPD) receiving triple or double inhaled maintenance therapy, and having had 1 or more documented COPD exacerbations in the 12 months prior to Visit 1. Subjects will receive CM512, or placebo, administered via subcutaneous injection at the study site, over a 52 week treatment period. The study also includes a post-treatment follow-up period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 40 to ≤ 80 years old

  * BMI ≥ 18.0 kg/(m*m)
  * COPD diagnosis≥1 year
  * Post-BD FEV1 ≥ 30% and < 80%, FEV1/FVC <0.70 at screening
  * Triple (LABA+LAMA+ICS) or dual inhaled (LABA+LAMA or LABA+ICS) COPD therapy ≥3 months prior to V1
* 2 moderate or ≥1 severe COPD exacerbations in the prior year

  * CAT ≥10 at screening
  * Former or current smokers ≥10 pack-years

Exclusion Criteria:

* Clinically important pulmonary disease other than COPD, as judged by the Investigator (including current or historic asthma diagnosis).
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable.
* Treatment with oxygen of more than 15 hours per day.
* Pregnant or breastfeeding.
* The chest/lungs with pathology that precludes the patient's ability to complete the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2028-03-17 (Estimated); Study Completion 2028-03-17 (Estimated)

PRIMARY OUTCOMES:
Annualised rate of moderate or severe COPD exacerbations | Baseline up to 52 weeks
  The annualised moderate or severe COPD exacerbation rate (based on exacerbations reported by the investigator) up to 52 weeks treatment period compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Jinfu Xu, Principal Investigator — Huadong Hospital